CLINICAL TRIAL: NCT07003165
Title: Research on a New Intelligent Mobile Screening and Diagnosis Pattern for Ocular Diseases
Status: Not yet recruiting | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025KYPJ044
Record Dates: First submitted 2025-05-25; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Ophthalmic Diseases (Specific Types Not Restricted); Cataract; Refraction Error; Diabetic Retinopathy (DR); Age Related Macular Degeneration (ARMD)
MeSH Terms: conditions — Cataract; Refractive Errors; Diabetic Retinopathy; Macular Degeneration

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intelligent Mobile Group: Participants were first screened for mobile eye health risk classification, and those who met the requirements were further screened by eye examination on the mobile clinic and suspected cases were recommended to be referred to higher level hospitals for consultation, and corresponding data were collected at different visit points.

SUMMARY:
The global distribution of primary ophthalmic medical resources is uneven, and the traditional eye disease screening model has problems such as low efficiency, high cost and limited coverage. With the development of artificial intelligence and other technologies, it provides technical support for the construction of intelligent mobile screening model for eye diseases. The investigator's team has developed the 5G intelligent ophthalmic vehicle and served tens of thousands of people in 108 cities nationwide, initially verifying the feasibility of the new intelligent mobile screening model. However, the application effect, acceptance and influencing factors of this model in different regions are not clear, and there is a lack of economic benefit analysis based on real-world data. In this study, the investigators will conduct a cross-sectional study of large-scale population screening for blinding eye diseases in grassroots areas through the smart mobile screening model, focusing on the screening effectiveness and cost-effectiveness of the smart mobile screening model, integrating real-world multimodal eye health data, developing multiple smart screening analysis models, and exploring its adaptability and direction of improvement in grassroots areas.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 7 years
* Voluntary informed consent

Exclusion Criteria:

-Inability to complete the required examinations with the help of others due to old age, infirmity, poor general condition, etc.

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: community sample or primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Cost-effectiveness | Baseline,6months,12months
  Incremental Cost per True Positive Case Detected

SECONDARY OUTCOMES:
Eye disease detection rate | Baseline,6months,12months
Accuracy of multiple intelligent screening analysis models | Baseline
Screening participation rate | baseline